CLINICAL TRIAL: NCT07388498
Title: A Phase 3, Multicenter, Double-blind, Randomized Controlled Study Evaluating the Efficacy and Safety of Pegloticase Administered by Subcutaneous Injection Compared With Pegloticase Administered by Intravenous Injection, Both Administered Concurrently With Methotrexate Weekly, in Participants With Uncontrolled Gout
Brief Title: A Double-blind, Randomized Controlled Trial to Investigate the Efficacy, Safety, and Pharmacokinetics of Pegloticase Administration Via Subcutaneous and Intravenous Routes Both With Methotrexate in Participants With Uncontrolled Gout
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230219
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Uncontrolled Gout
Keywords: Uncontrolled Gout; Pegloticase; KRYSTEXXA; Kadence
MeSH Terms: interventions — Pegloticase; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegloticase SC with MTX (Experimental): Participants will receive pegloticase SC every two weeks with MTX.
  Interventions: Drug: Pegloticase; Drug: Methotrexate
- Pegloticase IV with MTX (Experimental): Participants will receive pegloticase IV every two weeks with MTX.
  Interventions: Drug: Pegloticase; Drug: Methotrexate

INTERVENTIONS:
Drug: Pegloticase — Participants will receive pegloticase either SC or IV.
  Other Names: KRYSTEXXA
Drug: Methotrexate — MTX will be administered orally.
  Other Names: MTX

SUMMARY:
The primary objective of this trial is to evaluate the effect of pegloticase 18 mg subcutaneously (SC) every two weeks with methotrexate (MTX) versus pegloticase 8 mg intravenously (IV) every two weeks with MTX on the response rate during Month 6, as measured by the sustained normalization of serum uric acid (sUA) to < 6 mg/dL for at least 80% of the time during Month 6.

ELIGIBILITY:
Inclusion Criteria

* Participant has provided informed consent before initiation of any trial-specific activities/procedures.
* Age ≥ 18 years or ≥ legal age within the country if it is older than 18 years.
* Participants willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.
* Participants with uncontrolled gout, as meeting the protocol defined criteria.

Exclusion Criteria

* Glucose-6-phosphate dehydrogenase deficiency (tested at the screening visit).
* Liver transaminase levels (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) > 1.25 x upper limit of normal (ULN) or albumin < the lower limit of normal (LLN) at the screening visit.
* Uncontrolled diabetes mellitus and/or hemoglobin A1c (HbA1c) > 8%.
* Known intolerance to MTX.
* Participant received prior treatment with pegloticase, another recombinant uricase (ie, rasburicase or pegadricase), or concomitant therapy with a polyethylene glycol (PEG)-conjugated drug.
* A known intolerance to all protocol standard gout flare prophylaxis regimens (ie, participant must be able to tolerate at least 1 of the following: colchicine and/or non-steroidal anti-inflammatory drug and/or low-dose prednisone ≤ 10 mg/day or equivalent dose of other corticosteroid).
* Chronic renal impairment defined as estimated glomerular filtration rate (eGFR) based on Modification of Diet in Renal Disease (MDRD) calculations < 40 mL/min/1.73 m^2 or currently on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-02-19 (Estimated); Primary Completion 2028-05-23 (Estimated); Study Completion 2028-07-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Month 6 Response at Weeks 20, 21, 22, 23, and 24 | Month 6 (Weeks 20, 21, 22, 23, and 24)
  Defined as Achieving and Maintaining sUA < 6 mg/dL for at Least 80% of the Time During Month 6.

SECONDARY OUTCOMES:
Number of Participants With Serious Injection Site Reactions Through Week 48 | Up to Week 48
Number of Participants With Serious Adjudicated Infusion Reactions (Including Adjudicated Anaphylaxis) Through Week 48 | Up to Week 48
Number of Participants With Adjudicated Anaphylaxis Through Week 48 | Up to Week 48
Serum Concentrations of Pegloticase Following SC and IV Administration | Up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- D and H National Research Centers, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this trial will be considered beginning 18 months after the trial has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this trial.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen trial/trials in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com